CLINICAL TRIAL: NCT04336800
Title: Multi-Parametric MRI Assessment of the Liver in Diabetic Volunteers (Partners Registry)
Status: Completed | Type: Observational
Sponsor: Perspectum (Industry)
Responsible Party: Sponsor
Other Study IDs: EC-248
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2
Keywords: NASH; Fatty Liver; Livermultiscan
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2; Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: LiverMultiscan — The LiverMultiscan is a quick 15 min, contrast free scan that non-invasively provides three metrics of liver health namely liver fat, iron and fibro-inflammation

SUMMARY:
To build a registry of diabetic volunteers by inviting them to get a LiverMultiScan and collecting their contact information to seek interest in participating in future research studies.

DETAILED DESCRIPTION:
Perspectum's LiverMultiScan is a quantitative multiparametric MRI method, FDA-cleared and CE-marked, that is used to detect and stage early liver disease.It is already widely used internally in both research and within the clinical setting. LiverMultiScan has been adopted as the only liver scan in whole-population long term studies. The LiverMultiScan is more cost efficient, short in duration(<15mins), non-invasive and safe(no IV or oral contrast required, no ionizing radiation and no venipuncture).

This is a registry where there will be no intervention to the standard of care. Registry volunteers will be required to attend a single visit that will involve having a multi-parametric MRI at no cost to them. In addition, the investigators will collect contact information of the volunteers including their email address, phone number and home address so that they can be contacted to discuss possible participation in future studies which may be sponsored by Perspectum or third parties, such as pharmaceutical companies.The volunteer's personal information shall never be shared with these third parties. Additionally, the contact information of the volunteers' medical providers shall also be collected so that the LiverMultiScan reports can be delivered to them.

ELIGIBILITY:
Inclusion Criteria:

* Male or female diabetic volunteers aged 18 years and over who are willing and able to give informed consent for participation in the registry.

Exclusion Criteria:

* The volunteer may not enter the registry if they have any contraindication to magnetic resonance imaging (standard MR exclusion criteria at the imaging center including pregnancy, extensive tattoos, pacemaker, shrapnel injury, severe claustrophobia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic volunteers who are willing to get an MRI scan for the assessment of their liver
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
To build a registry of diabetic volunteers by inviting them to get a LiverMultiScanand collecting their contact information to seek interest in participating in future studies. | 12 months

SECONDARY OUTCOMES:
To use multi-parametric MRI (LiverMultiScan) of the liver to assess liver health | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Partners Imaging Centers, Sarasota, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided